CLINICAL TRIAL: NCT05910996
Title: Prediction of Conversion From Vv-ECMO to Va-ECMO in COVID-19 Patients
Acronym: ECMOPred-vvva
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECMOPred-vvva
Record Dates: First submitted 2023-06-15; First posted 2023-06-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: ARDS Due to Disease Caused by SARS Co-V-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conversion from vv-ECMO to va-ECMO Positive
  Interventions: Procedure: Conversion from vv-ECMO to va-ECMO
- Conversion from vv-ECMO to va-ECMO Negative

INTERVENTIONS:
Procedure: Conversion from vv-ECMO to va-ECMO — Conversion from vv-ECMO to va-ECMO
  Groups: Conversion from vv-ECMO to va-ECMO Positive

SUMMARY:
In December 2019, cases of a novel lung disease, later referred to as COVID-19, were first reported in China. The virus SARS-CoV-2 was identified as the causative agent. Due to the sharp increase in the number of cases worldwide, a pandemic outbreak was declared by WHO in March 2020.

The infection presents with a broad clinical spectrum. Frequently, there is respiratory infection with fever (80%), dry cough (56%), fatigue (22%), and muscle pain (7%), but completely asymptomatic infection is also possible. Severe courses may be associated with pneumonia resulting in acute respiratory distress syndrome (ARDS) requiring intensive care.

In the context of intensive care therapy, it is sometimes necessary to use extracorporeal organ replacement procedures due to increasing lung failure. In this context, extracorporeal membrane oxygenation (ECMO) was used during the pandemic. With this procedure it is possible to replace on the one hand the oxygenation and ventilation function of the lung and on the other hand additionally the pumping function of the heart, if configured appropriately. The switch from venovenous (vv) configuration, with which only lung function is replaced, to venoarterial (va) configuration (lung function and heart function are replaced) is made in cases of intensive care necessity, e.g., increasing decompensation of heart failure.

Heart failure manifests itself, among other things, through insufficient pumping function of the heart muscle. This results in an undersupply of peripheral tissues with arterial blood, leading to increased anaerobic glycolysis. Lactate and B-type natriuretic peptide (BNP) are used as surrogate parameters of this undersupply. Increased oxygen depletion from oxygen available in arterial blood is detected by the surrogate parameter central venous oxygen saturation (ScvO2).

In addition to ECMO, drug interventions are also used to improve cardiorespiratory performance at various doses. As described by Suwalski et al, there may be a relationship between this drug therapy and conversion from vv to va ECMO.

Currently, few studies exist on conversion from vv-ECMO to va-ECMO. In this regard, Suwalski et al. describe a population that experienced any ECMO therapy for a maximum period of 16.5 ± 10.0 days, with the group with conversion receiving 17.8 ± 10.5 days of therapy and the group without conversion receiving 16.4 ± 9.4 days. The need for conversion to va-ECMO requires additional expertise that is not readily available despite acute intensive care transport readiness. It is likely that by predicting the need for conversion, early logistical planning for transfer to an appropriate center with experience and equipment can occur, or if transfer is not necessary, staffing and equipment preparation can occur earlier and more safely. As described by Falk et al, planned and prepared conversion can also be expected to have an impact on patient* survival.

The aim of this retrospective, exploratory data analysis is to predict conversion before placement of vv-ECMO within 30 days from ICU care from vv-ECMO to va-ECMO in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients aged 18 years or older that were treated in intensive care at the study center between 2019-12-01 and 2023-04-15.

Exclusion Criteria:

* Patients in which ECMO therapy was started outside of the study center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Confusion Matrix | 2019-12-01 to 2023-07-01
  Confusion Matrix for Classification of Conversion from vv-ECMO to va-ECMO

SECONDARY OUTCOMES:
Mortality | 2019-12-01 to 2023-07-01
  7, 14, and 30 Day-In Hospital Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No